CLINICAL TRIAL: NCT01868581
Title: A Randomised, Single Centre, Double-blind, Two-period Crossover, Glucose Clamp Trial to Test for Bioequivalence Between Two Insulin 454 Formulations, With or Without Buffer, and Between Two SIAC Formulations, With or Without Buffer, in Healthy Male Subjects
Brief Title: Bioequivalence Between Two Explorative Insulin Degludec Formulations and Between Two Explorative IDegAsp Formulations in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN5401-1985; 2008-000097-20 (EudraCT Number)
Record Dates: First submitted 2013-05-30; First posted 2013-06-04 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — insulin degludec; insulin degludec, insulin aspart drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- insulin degludec (Experimental)
  Interventions: Drug: insulin degludec
- IDegAsp (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart

INTERVENTIONS:
Drug: insulin degludec — Each subject will be allocated to 2 single injections of trial product on 2 separate dosing visits, administered subcutaneously (s.c., under the skin).
  Arms: insulin degludec
Drug: insulin degludec/insulin aspart — Each subject will be allocated to 2 single injections of trial product on 2 separate dosing visits, administered subcutaneously (s.c., under the skin).
  Arms: IDegAsp

SUMMARY:
This trial is conducted i Europe. The aim of this trial is to test for bioequivalence between two explorative formulations of insulin degludec (insulin 454) and between two explorative insulin degludec/insulin aspart (IDegAsp - formerly SIAC) formulations, all with or without buffer, in healthy male subjects. The investigated formulations are explorative, not similar to the proposed commercial formulation.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial related activities are any procedure that would not have been performed during the normal management of the subject
* Considered generally healthy upon completion of medical history and physical examination as judged by the Investigator
* Body mass index (BMI) between 18.0 and 27.0 kg/m^2 (inclusive)
* Fasting plasma glucose below or equal to 6 mmol/L
* Sexually active and non-sterilised participants must be informed that they and their partner must use a safe method of contraception during sexual intercourse (risk of pregnancy must be lower than 1%), e.g. implants, injections, combined oral contraceptives or hormonal intrauterinedevice or be willing to refrain from having sexual intercourse from the beginning of the study until up to three months after the conclusion of the study. This serves to exclude the possibilityof a pregnancy through sperm that could have been damaged by the study medication

Exclusion Criteria:

* A history of any illness that, in the opinion of the investigator, might confound the results of the trial or pose risk in administering the trial product to the subject
* Known or suspected allergy to trial products or related products
* Subject who has participated in any other trials involving investigational products within the last 3 months prior to first dosing

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2008-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Area under the serum insulin degludec concentration-time curve (for insulin degludec) | 0-120 hours after dosing
Maximum serum insulin degludec concentration (Cmax) (for insulin degludec) | 0-120 hours after dosing
Area under the serum insulin aspart concentration-time curve (for IDegAsp) | 0-10 hours after dosing
Maximum serum insulin aspart concentration (Cmax) (for IDegAsp) | 0-10 hours after dosing
Area under the serum insulin degludec concentration-time curve (for IDegAsp) | 0-120 hours after dosing
Maximum serum insulin degludec concentration (Cmax) (for IDegAsp) | 0-120 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Neuss, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com